CLINICAL TRIAL: NCT00905125
Title: A Randomized, Double-Blind Trial on the Safety and Immunogenicity of Inactivated Trivalent Influenza Vaccine in Pregnant Women
Brief Title: Influenza Vaccine in Pregnant Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 09-0033; N01AI80002C
Record Dates: First submitted 2009-05-18; First posted 2009-05-20 (Estimated); Results first posted 2011-04-06 (Estimated); Last update posted 2012-06-13 (Estimated); Status verified 2010-03

CONDITIONS: Influenza
Keywords: influenza, trivalent, vaccine, pregnant women
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines; fluarix

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Arm 2, Fluarix® (Experimental): Single 0.5 mL intramuscular injection of Fluarix®.
  Interventions: Biological: Fluarix®
- Arm 1, Fluzone® (Experimental): Single 0.5 mL intramuscular injection of Fluzone®.
  Interventions: Biological: Fluzone®

INTERVENTIONS:
Biological: Fluzone® — Single 0.5 mL injection of the 2008-2009 seasonal inactivated trivalent influenza vaccine administered intramuscularly in the deltoid. Fluzone® does not contain thimerosal.
  Arms: Arm 1, Fluzone®
Biological: Fluarix® — Single 0.5 mL injection of the 2008-2009 seasonal inactivated trivalent influenza vaccine administered intramuscularly in the deltoid. Fluarix® contains less than 1 microgram (trace or a very small amount) thimerosal per shot.
  Arms: Arm 2, Fluarix®

SUMMARY:
In pregnant women, flu may cause complications like pneumonia (infection of the lungs) or hospitalization. In the United States (US) it is recommend that all women get flu vaccine if they are going to be pregnant or deliver during the flu season but only a few studies have measured a pregnant woman's immune response (the body's defense against the flu) after getting the flu vaccine. About 200, 18-39 year old, inclusive, pregnant women in their second or third trimester (from 14 weeks of gestation to term, inclusive) will be enrolled in this US based study. Participation will be about 8 months in duration. Women will be randomized (assigned by chance) to receive either Fluzone® or Fluarix®. Blood collection will occur on Day 0 and 28 days post vaccination.

DETAILED DESCRIPTION:
Influenza is a significant cause of morbidity and mortality in the United States (US), resulting in an average of 226,000 hospitalizations and 36,000 deaths each year. Pregnant women and infants are at an increased risk for the complications of influenza. Severe disease, emergency department visits and hospitalizations occur frequently in pregnant women and infants which are considered high risk populations. In the US, routine vaccination with inactivated trivalent influenza vaccine (TIV) is recommended for pregnant women or those who deliver during the influenza season. Few studies exist on the safety and immunogenicity of administration of seasonal inactivated TIV despite long-standing recommendations. Although influenza vaccination has been recommended during pregnancy, the rates of immunization remain low, at about 13 percent. This is a multi-site randomized, double-blind clinical trial in 200 ambulatory, medically stable 18-39 year old, inclusive, pregnant women in their second or third trimester of pregnancy (from 14 weeks of gestation to term, inclusive). Study subjects will be randomized 1:1 to receive one dose of a 2008-2009 seasonal inactivated TIV, either Fluzone® or Fluarix® (100 pregnant women per vaccine group). Once enrolled, a blood sample will be collected and each subject will receive a single 0.5 mL dose of a 2008-2009 seasonal inactivated TIV, either Fluzone® or Fluarix®. The vaccination will occur on Day 0. Subjects will be observed for approximately 15 minutes after vaccination. All subjects will maintain a memory aid recording oral temperature, and systemic and local adverse events (AEs) for 7 days after each vaccination. Subjects will be encouraged to take their temperature around the same time each day. Subjects will have a phone call on Day 2 for review of memory aid, concomitant medication assessment, and assessment of AEs. Subjects will have a phone call on Day 8 for AE assessment, concomitant medication assessment and review of memory aid. At approximately Day 28 after the vaccination, subjects will return to the clinic for immunogenicity blood sample collection, concomitant medication assessment, and assessment of any AEs. A targeted physical exam will be conducted, if indicated. At approximately Day 180 or 6 months after vaccination, subjects will have a phone call for assessment for any serious adverse events (SAEs). Unsolicited non-serious AE data will be captured Day 0 through Day 28. Maternal SAE data will be captured throughout the study period (Day 0 through Day 180, approximately 6 months after dose of vaccine). Maternal and infant SAE data will be collected when obtaining data on pregnancy outcome. Serum for immunogenicity evaluations will be obtained prior to the dose of vaccine (at Day 0); and one month after vaccination (at Day 28). Pregnancy outcome data will be captured by a review of medical records and a phone call to the subject. Data include any complications during labor and delivery for both the mother as well as the neonate, to include premature delivery or delivery by emergency cesarean section. Neonatal assessments will include but not be limited to gestational age, birth weight, Apgar scores, congenital abnormalities, infection, hematological and metabolic complications, admission to nursery or Neonatal Intensive Care Unit and the need for respiratory support. Blood samples collected will be tested in a central laboratory for the levels of hemagglutination inhibition (HAI) and microneutralization (MN) antibodies.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant female between the ages of 18 and 39 years, inclusive.
* Is from 14 weeks of gestation to term, inclusive.
* Is in good health, as determined by vital signs (heart rate <100 bpm; blood pressure: systolic <140 mm Hg; diastolic less than or equal to 90 mm Hg; oral temperature <100.0 degrees Fahrenheit), medical history to ensure stable medical condition and a targeted physical examination based on medical history (if indicated). A stable medical condition is defined as health outcomes of the specific disease are considered to be within acceptable limits in the last 3 months.
* Able to understand and comply with planned study procedures.
* Provides written informed consent prior to initiation of any study procedures.
* Agrees to sign medical release for herself and her infant(s) to allow study staff to gather pregnancy outcome data, if needed per clinical site policy.

Exclusion Criteria:

* Receipt of the 2008-2009 seasonal influenza vaccine [trivalent inactivated vaccine (TIV) or Flumist] prior to enrollment into the study.
* Has a known allergy to eggs, egg proteins, latex allergy or allergy to other components in the vaccines (i.e. formaldehyde, polyethylene glycol p-isooctylphenyl ether, sucrose, gelatin, polysorbate 80).
* Has a history of severe reactions following immunization with contemporary influenza virus vaccines.
* Has received any other licensed vaccines within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) prior to vaccination in this study or expects to receive a licensed product prior to Visit 4 (Day 28 visit) (except for inactivated influenza vaccine which may be received 2 weeks post vaccination with study product). Measles, mumps, rubella vaccine is permitted post-partum.
* Has a moderate-to-severe acute illness and/or an oral temperature greater than or equal to 100.0 degrees Fahrenheit, within 72 hours prior to vaccination. (This may result in a temporary delay of vaccination).
* Immunosuppression as a result of an underlying illness or treatment, or use of anti-cancer chemotherapy or radiation therapy within the preceding 36 months.
* Has an active neoplastic disease, a history of any hematologic malignancy, current bleeding disorder, or taking anticoagulants.
* Long term use of oral or parenteral steroids, high-dose inhaled steroids (>800 mcg/day of beclomethasone dipropionate or equivalent) within the preceding 6 months (nasal and topical steroids are allowed) or has received steroids for treatment of pre-term labor during this pregnancy.
* Has a history of receiving immunoglobulin or other blood product (with exception of Rhogam) within the 3 months prior to vaccination in this study.
* Has a diagnosis of a current and uncontrolled major psychiatric disorder.
* The subject is receiving listed psychiatric drugs (aripiprazole, clozapine, ziprasidone, haloperidol, molindone, loxapine, thioridazine, thiothixene, pimozide, fluphenazine, risperidone, mesoridazine, quetiapine, trifluoperazine, trifluopromazine, chlorprothixene, chlorpromazine, perphenazine, olanzapine, carbamazepine, divalproex sodium, lithium carbonate or lithium citrate). Subjects who are receiving an antidepressant drug and are stable for at least 3 months prior to enrollment without decompensating are allowed enrollment into the study.
* Known active human immunodeficiency virus, hepatitis B, or hepatitis C infection.
* History of alcohol or drug abuse in the 1 year prior to enrollment.
* Has a history of Guillain-Barré syndrome.
* Has a seizure disorder or is on an anti-seizure medication for a seizure disorder.
* Has received an experimental/investigational agent (vaccine, drug, biologic, device, blood product, or medication) during this pregnancy prior to enrollment, or expects to receive an experimental/investigational agent prior to Visit 4 (Day 28 visit).
* Has an acute or chronic medical condition that, in the opinion of the investigator would interfere with the evaluation of responses (this includes, but is not limited to: known chronic liver disease, significant renal disease, transplant recipients, uncontrolled diabetes, juvenile diabetes (Type 1) or advanced diabetes with renal and eye disease; diabetes controlled by diet or oral agents is acceptable).
* Has any condition that would, in the opinion of the site investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2009-06; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Emory University School of Medicine - Gynecology and Obstetrics, Atlanta, Georgia
  - University of Iowa, Iowa City, Iowa
  - University of Maryland Baltimore, Baltimore, Maryland
  - Mayo Clinic, Rochester - Vaccine Research Group, Rochester, Minnesota
  - Saint Louis University, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - Vanderbilt University, Nashville, Tennessee
  - Baylor College of Medicine - Molecular Virology and Microbiology, Houston, Texas
  - Group Health Cooperative, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment began on 11JUN2009 and was closed on 03SEP2009 due to the availability of the 2009-2010 seasonal Influenza vaccine and onset of Influenza season.
Groups:
- Fluzone®: Single 0.5 mL intramuscular injection of Fluzone®
- Fluarix®: Single 0.5 mL intramuscular injection of Fluarix®
Period: Overall Study
Arm/Group | Fluzone® | Fluarix®
Started | 46 | 56
Completed | 42 | 53
Not Completed | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluzone® | Fluarix® | Total
Number analyzed (Participants) | 46 | 56 | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 46 | 56 | 102
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 28.0 (5.9) | 28.4 (5.0) | 28.2 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 56 | 102
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 46 | 56 | 102

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Serum Hemagglutination Inhibition Assay (HAI) Antibody Titer Greater Than or Equal to 40 Against Each Antigen Included in the 2008-2009 Seasonal Inactivated Trivalent Influenza Vaccine (TIV)
Description: Blood was collected for HAI assay at Day 0 prior to vaccination and again at 28 days following vaccination. The HAI assay was conducted with the three antigens in the 2008-2009 seasonal inactivated TIV: Influenza B antigen, H1N1 antigen, and H3N2 antigen.
Time Frame: Day 0 prior to and Day 28 after receiving single dose.
Population: Participants are included in this ITT analysis if blood was collected at both timepoints. One participant was excluded because the baseline blood draw was done after vaccination.
Measure: Number; unit: Participants
Arm/Group | Fluzone® | Fluarix®
Number analyzed (Participants) | 45 | 55
Participants
  Influenza B antigen, Day 0 | 4 | 3
  Influenza B antigen, Day 28 | 35 | 33
  Influenza H1N1 antigen, Day 0 | 7 | 7
  Influenza H1N1 antigen, Day 28 | 43 | 47
  Influenza H3N2 antigen, Day 0 | 14 | 22
  Influenza H3N2 antigen, Day 28 | 42 | 51

2. Primary Outcome: Number of Participants Reporting Maternal Complications of Pregnancy, Labor and Delivery.
Description: Participants were contacted after delivery, and medical records reviewed, to collect complications experienced during pregnancy, labor and delivery. The data collection process followed a prospectively-defined list of complications reported for this outcome measure, some of which may have also been reported as serious adverse events if otherwise meeting those requirements.
Time Frame: At time of delivery.
Population: All participants from whom outcome data were collected are included in the ITT safety population for this outcome measure.
Measure: Number; unit: Participants
Arm/Group | Fluzone® | Fluarix®
Number analyzed (Participants) | 45 | 55
Participants
  Stillborn | 1 | 1
  Miscarriage | 1 | 0
  Gestational diabetes | 2 | 4
  Polyhydramnios | 1 | 0
  Oligohydramnios | 5 | 2
  Pregnancy induced hypertension | 2 | 4
  Pre-eclampsia | 1 | 6
  Eclampsia | 0 | 0
  Fetal distress | 1 | 5
  Abruptio placenta | 1 | 0
  Chorioamnionitis | 2 | 3
  Fever greater than 100.4 degrees Fahrenheit | 4 | 5
  Anaphylaxis | 0 | 0
  Antibiotics prior to delivery | 18 | 21
  Fetal abnormalities detected during pregnancy | 2 | 2
  Assisted vaginal delivery | 3 | 3
  Non-elective Cesarean section | 7 | 9
  Abnormal amniotic fluid | 13 | 11
  Postpartum fever | 3 | 1
  Postpartum endometritis | 1 | 0
  Postpartum bleeding | 2 | 2
  Postpartum bacteremia | 0 | 0

3. Primary Outcome: Number of Participants Reporting Neonatal Complications.
Description: Participants were contacted after delivery, and medical records reviewed, to collect neonatal complications. The data collection process followed a prospectively-defined list of complications reported for this outcome measure, some of which may have also been reported as serious adverse events if otherwise meeting those requirements.
Time Frame: At time of delivery.
Population: All live births are included in this outcome measure, which excludes three participants whose pregnancies ended in miscarriage or stillbirth (reported as maternal complications). Three participants gave birth to twins, who are each counted separately.
Measure: Number; unit: Participants
Arm/Group | Fluzone® | Fluarix®
Number analyzed (Participants) | 44 | 56
Participants
  Pre-term (less than 37 weeks) | 3 | 4
  Large for gestational age | 4 | 9
  Small for gestational age | 3 | 2
  Abnormal infant exam | 8 | 11
  Congenital abnormalities | 4 | 2
  Hematological complications | 0 | 5
  Infection | 0 | 1
  Sepsis | 0 | 0
  Meningitis | 0 | 0
  Metabolic complications | 0 | 0
  Respiratory complications | 7 | 4
  Respiratory support used | 5 | 4
  Fever 100.4 degrees Fahrenheit or greater | 1 | 0
  Admission to special nursery/intensive care | 7 | 3

4. Primary Outcome: Number of Participants Reporting Serious Adverse Events (SAE)
Description: Serious adverse events included any untoward medical occurrence that resulted in death of the mother, fetus or infant; was life threatening to mother, fetus or infant; was a persistent/significant disability/incapacity; required in-patient hospitalization or prolongation thereof; was a congenital anomaly/birth defect in fetus or infant; or may have jeopardized the mother, fetus or infant, or required intervention to prevent one of the outcomes. All events are included regardless of association to vaccination.
Time Frame: Through 6 months post vaccination.
Population: All participants are included in the ITT safety population for this outcome measure.
Measure: Number; unit: Participants
Arm/Group | Fluzone® | Fluarix®
Number analyzed (Participants) | 46 | 56
Participants | 8 | 13

5. Primary Outcome: Number of Participants Reporting Unsolicited Non-serious Adverse Events Considered Associated With Vaccination
Description: Unsolicited non-serious adverse events were collected from participants at follow up contacts, either by phone or in clinic, through 28 days after vaccination. Association to vaccination was determined by a clinician licensed to make a medical diagnosis and listed on the site's Federal Drug Administration's Form 1572.
Time Frame: Day 0 through Day 28 post vaccination.
Population: All participants are included in the ITT safety population for this outcome measure.
Measure: Number; unit: Participants
Arm/Group | Fluzone® | Fluarix®
Number analyzed (Participants) | 46 | 56
Participants | 0 | 3

6. Primary Outcome: Number of Participants Reporting Solicited Injection Site Reactions at Each Severity Based on the Functional Grading Scale
Description: Participants recorded a daily maximum severity at which local reactions of pain, tenderness and swelling were experienced. Mild reactions had no interference with daily activities, moderate reactions interfered with daily activity, and severe reactions were defined as preventing daily activity. Participants are reported at the highest severity experienced across the 8 days.
Time Frame: Days 0-7 after vaccination.
Population: All participants are included in the ITT safety population for this outcome measure.
Measure: Number; unit: Participants
Arm/Group | Fluzone® | Fluarix®
Number analyzed (Participants) | 46 | 56
Participants
  Mild pain | 14 | 22
  Moderate pain | 4 | 1
  Severe pain | 0 | 0
  Mild tenderness | 34 | 39
  Moderate tenderness | 4 | 2
  Severe tenderness | 0 | 0
  Mild swelling | 3 | 3
  Moderate swelling | 0 | 0
  Severe swelling | 0 | 0

7. Secondary Outcome: Number of Participants With a Serum Microneutralization Antibody Titer of Greater Than or Equal to 40 Against Each Antigen in the 2008-2009 TIV
Description: Blood was collected for microneutralization assay at Day 0 prior to vaccination and again at 28 days following vaccination. The microneutralization assay was to be conducted with the three antigens in the 2008-2009 seasonal inactivated TIV: Influenza B antigen, H1N1 antigen, and H3N2 antigen.
Time Frame: Day 0 prior to and Day 28 after receiving a single dose.
Population: Microneutralization assays were deemed not necessary by the sponsor and conduct of these assays is not planned.
Measure: Number; unit: Participants
Arm/Group | Fluzone® | Fluarix®
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Number of Participants With a Four-fold or Greater Rise in Microneutralization Antibody Titer Against Each Antigen in the 2008-2009 TIV
Description: Blood was collected for microneutralization assay at Day 0 prior to vaccination and again at 28 days following vaccination. The microneutralization assay was to be conducted with the three antigens in the 2008-2009 seasonal inactivated TIV: Influenza B antigen, H1N1 antigen, and H3N2 antigen. The threshold of a four-fold increase in titer would be met if the Day 0 titer was less than 10 (the assay's lowest level of detection) and the Day 28 titer was 40 or greater, or the Day 0 titer was greater than or equal to 10, and the Day 28 titer was an increase by four-fold or more.
Time Frame: Day 0 prior to and Day 28 receiving a single dose.
Population: Microneutralization assays were deemed not necessary by the sponsor and conduct of these assays is not planned.
Measure: Number; unit: Participants
Arm/Group | Fluzone® | Fluarix®
Number analyzed (Participants) | 0 | 0

9. Primary Outcome: Number of Participants Reporting Measured Injection Site Reactions of Swelling and Redness at Each Grade
Description: Participants recorded a daily measured value of swelling and redness, if present. The protocol defined grading of small, medium and large, with small as less than 20 mm, medium as 20-50 mm and large as greater than 50 mm. Participants are counted at the largest measured grade experienced across the 8 day period after vaccination.
Time Frame: Days 0-7 after vaccination.
Population: All participants are included in the ITT safety population for this outcome measure.
Measure: Number; unit: Participants
Arm/Group | Fluzone® | Fluarix®
Number analyzed (Participants) | 46 | 56
Participants
  Small swelling | 2 | 3
  Medium swelling | 2 | 1
  Large swelling | 0 | 0
  Small redness | 4 | 7
  Medium redness | 3 | 1
  Large redness | 0 | 0

10. Primary Outcome: Number of Participants Reporting Solicited Systemic Symptoms at Each Severity Based on the Functional Grading Scale
Description: Participants recorded a daily maximum severity at which systemic symptoms of feverishness, malaise, myalgia, headache and nausea were experienced. Mild reactions had no interference with daily activities, moderate reactions interfered with daily activity, and severe reactions were defined as preventing daily activity. Participants are reported at the highest severity experienced across the 8 days.
Time Frame: Days 0-7 after vaccination.
Population: All participants are included in the ITT safety population for this outcome measure.
Measure: Number; unit: Participants
Arm/Group | Fluzone® | Fluarix®
Number analyzed (Participants) | 46 | 56
Participants
  Mild feverishness | 5 | 2
  Moderate feverishness | 0 | 0
  Severe feverishness | 0 | 0
  Mild malaise | 11 | 15
  Moderate malaise | 7 | 10
  Severe malaise | 1 | 0
  Mild myalgia | 6 | 6
  Moderate myalgia | 3 | 3
  Severe myalgia | 0 | 0
  Mild headache | 10 | 7
  Moderate headache | 6 | 0
  Severe headache | 0 | 0
  Mild nausea | 7 | 6
  Moderate nausea | 1 | 6
  Severe nausea | 0 | 0

11. Primary Outcome: Number of Participants Reporting Fever Based on the Protocol-defined Grading Scale for Oral Temperature
Description: Participants recorded a daily oral temperature on a memory aid for 8 days (Days 0-7) after vaccination. The protocol defined mild fever as oral temperatures 37.8 to less than 38 degree Celsius, moderate fever as 38 to less than 39 degrees Celsius and severe fever as oral temperatures of 39 degrees Celsius or higher. Participants are reported at the highest severity experienced across the 8 days.
Time Frame: Days 0-7 after vaccination.
Population: All participants are included in the ITT safety population for this outcome measure.
Measure: Number; unit: Participants
Arm/Group | Fluzone® | Fluarix®
Number analyzed (Participants) | 46 | 56
Participants
  Mild fever | 0 | 0
  Moderate fever | 0 | 0
  Severe fever | 0 | 0

12. Primary Outcome: Hemagglutination Inhibition Assay (HAI) Geometric Mean Titer (GMT) Against Each Antigen in the 2008-2009 Seasonal Influenza Trivalent Influenza Vaccine
Description: as for outcome 1
Time Frame: Day 0 prior to and Day 28 after receiving single dose.
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Titer
Arm/Group | Fluzone® | Fluarix®
Number analyzed (Participants) | 45 | 55
Titer
  Influenza B antigen, Day 0 | 10.8 [8.1 to 14.4] | 10.0 [8.1 to 12.5]
  Influenza B antigen, Day 28 | 67.5 [52.8 to 86.5] | 41.7 [33.5 to 52.0]
  Influenza H1N1 antigen, Day 0 | 11.7 [8.5 to 16.0] | 10.9 [8.6 to 13.7]
  Influenza H1N1 antigen, Day 28 | 126.0 [95.6 to 166.2] | 126.4 [92.3 to 173.2]
  Influenza H3N2 antigen, Day 0 | 20.2 [15.0 to 27.1] | 23.6 [17.7 to 31.6]
  Influenza H3N2 antigen, Day 28 | 206.3 [141.1 to 301.8] | 205.3 [151.0 to 279.2]

13. Secondary Outcome: Microneutralization Assay Geometric Mean Antibody Titers Against Each Antigen in the 2008-2009 TIV
Description: as for outcome 7
Time Frame: Day 0 prior to and Day 28 after receiving a single dose.
Population: Microneutralization assays were deemed not necessary by the sponsor and conduct of these assays is not planned.
Measure: Number; unit: Participants
Arm/Group | Fluzone® | Fluarix®
Number analyzed (Participants) | 0 | 0

14. Primary Outcome: Number of Participants With a Four-fold or Greater Rise in HAI Antibody Titer Against Each Antigen in the 2008-2009 Seasonal Influenza Trivalent Influenza Vaccine
Description: Blood was collected for HAI assay at Day 0 prior to vaccination and again at 28 days following vaccination. The HAI assay was conducted with the three antigens in the 2008-2009 seasonal inactivated TIV: Influenza B antigen, H1N1 antigen, and H3N2 antigen. A participant met the threshold of a four-fold increase in titer if the Day 0 titer was less than 10 (the assay's lowest level of detection) and the Day 28 titer was 40 or greater, or the Day 0 titer was greater than or equal to 10, and the Day 28 titer was an increase by four-fold or more.
Time Frame: Day 0 prior to and Day 28 receiving a single dose.
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Fluzone® | Fluarix®
Number analyzed (Participants) | 45 | 55
Participants
  Influenza B antigen | 25 | 24
  Influenza H1N1 antigen | 35 | 39
  Influenza H3N2 antigen | 35 | 40

ADVERSE EVENTS:
Time Frame: Solicited systemic symptoms and injection site reactions were collected for 7 days after vaccination. Unsolicited adverse events were collected for 28 days after vaccination. Serious adverse events were collected for 6 months after vaccination.
Arm/Group | Fluzone® | Fluarix®
Serious Adverse Events (participants affected / at risk) | 8/46 | 13/56
Other Adverse Events (participants affected / at risk) | 42/46 | 50/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluzone® (N=46) | Fluarix® (N=56)
Retained products of conception (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1)
HELLP syndrome (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1)
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Premature labour (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Polydactyly (Congenital, familial and genetic disorders) | 1 (1) | 1 (1)
Intra-uterine death (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Thyroid malformation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Caesarean section (Surgical and medical procedures) | 1 (1) | 2 (2)
Neonatal asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Foetal heart rate deceleration (Cardiac disorders) | 0 (0) | 1 (1)
Rhesus incompatibility (Immune system disorders) | 0 (0) | 1 (1)
Pilonidal cyst congenital (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Congenital anomaly (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Premature baby (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Congenital central nervous system anomaly (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluzone® (N=46) | Fluarix® (N=56)
Feeling hot (General disorders) | 5 (5) | 2 (2)
Malaise (General disorders) | 19 (19) | 25 (25)
Myalgia (Musculoskeletal and connective tissue disorders) | 9 (9) | 9 (9)
Headache (Nervous system disorders) | 16 (16) | 7 (7)
Nausea (Gastrointestinal disorders) | 8 (8) | 12 (12)
Injection site pain (General disorders) | 18 (18) | 23 (23)
Tenderness (General disorders) | 38 (38) | 41 (41) — Tenderness was solicited as a reaction at the vaccination site.
Injection site erythema (General disorders) | 7 (7) | 8 (8)
Injection site swelling (General disorders) | 4 (4) | 4 (4)

LIMITATIONS AND CAVEATS:
In September of 2009, the trial was closed to enrollment prior to accruing the intended 200 participants due to the availability of the 2009-2010 seasonal Influenza vaccine and onset of Influenza season.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less